CLINICAL TRIAL: NCT04013750
Title: Effect of Modified Constraint Induced Movement Therapy on Upper Extremity Functions of Stroke Patients With Right/Left Hemisphere Damage: Single Blind Randomized Controlled Trial
Brief Title: Effect of mCIMT on Upper Extremity Functions of Stroke Patients With Right/Left Hemiplegia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Cansin Medin Ceylan, assistant doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 415687
Record Dates: First submitted 2019-04-12; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Stroke Patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- left hemiplegia (Experimental): Patients in the left hemiplegia group had 10 sessions of constraint induced movement therapy as groups of 4, 5 days a week. Each patient had modified constraint induced movement therapy 1 hour a day with professional support and performed home program by themselves 3 hours a day. Patients' less affected hands were limited by the help of a glove %50 of the time they were awake
  Interventions: Other: Modified Constraint Induced Movement Therapy
- right hemiplegia (Experimental): Patients in the right hemiplegia group had 10 sessions of constraint induced movement therapy as groups of 4, 5 days a week. Each patient had modified constraint induced movement therapy 1 hour a day with professional support and performed home program by themselves 3 hours a day. Patients' less affected hands were limited by the help of a glove %50 of the time they were awake
  Interventions: Other: Modified Constraint Induced Movement Therapy
- control (No Intervention): 10 patients with right hemiplegia and 10 patients with left hemiplegia formed the control group and these patients were in line for inpatient rehabilitation programme.

INTERVENTIONS:
Other: Modified Constraint Induced Movement Therapy — constraint-induced movement therapy (CIMT) is characterized by the restraint of the less effected upper limb accompanied by the shaping and repetitive task-oriented training of more affected upper extremity.
  Arms: left hemiplegia; right hemiplegia

SUMMARY:
The investigators aimed To analyze effect of modified constraint induced movement therapy on upper extremity functions and quality of life of subacute and chronic phase stroke patients with right/left hemisphere damage. A total of 40 patients (20 patients with right hemiplegia and 20 patients with left hemiplegia) were enrolled in our prospective, randomized and controlled trial. Patients were randomized in to three groups. The first group consists of 10 right hemiplegia patients and the second group consists of 10 left hemiplegia patients. First and second group of patients had 10 sessions of constraint induced movement therapy as groups of 4, 5 days a week. Each patient had modified constraint induced movement therapy 1 hour a day with professional support and performed home program by themselves 3 hours a day. Patients' less affected hands were limited by the help of a glove %50 of the time they were awake. Patients were examined before treatment, just after treatment and 3 months after treatment using Box-Block Test, cubes lined, card turned and object gripped in 30 seconds, time it takes to grip and carry a water filled glass to their mouth and putting it back, Motor Activity Log (MAL), Stroke Impact Scale, Fugl-Meyer Motor Assessment Scale.

DETAILED DESCRIPTION:
For the rehabilitation of the paretic upper extremity, the use of constraint induced movement therapy and the use of modified constraint induced movement therapy are the most effective treatment strategies. The investigators aimed To analyze effect of modified constraint induced movement therapy on upper extremity functions and quality of life of subacute and chronic phase stroke patients with right/left hemisphere damage.

A total of 40 patients (20 patients with right hemiplegia and 20 patients with left hemiplegia) were enrolled in our prospective, randomized and controlled trial. Patients were randomized in to three groups. The first group consists of 10 right hemiplegia patients and the second group consists of 10 left hemiplegia patients. First and second group of patients had 10 sessions of constraint induced movement therapy as groups of 4, 5 days a week. Each patient had modified constraint induced movement therapy 1 hour a day with professional support and performed home program by themselves 3 hours a day. Patients' less affected hands were limited by the help of a glove %50 of the time they were awake. 10 patients with right hemiplegia and 10 patients with left hemiplegia formed the control group and these patients were in line for inpatient rehabilitation programme. Patients were examined before treatment, just after treatment and 3 months after treatment using Box-Block Test, cubes lined, card turned and object gripped in 30 seconds, time it takes to grip and carry a water filled glass to their mouth and putting it back, Motor Activity Log (MAL), Stroke Impact Scale, Fugl-Meyer Motor Assessment Scale. Wilcoxon Signed Ranks test and Friedman test were used for intragroup comparison of data and Kruskal-Wallis test was used to compare data between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients in subacute and chronic period (3 months after stroke)
* Modified Ashworth scale in the hemiplegic arm with 3 or more spasticity
* No pain in the hemiplegic arm
* MMSE 20 and above
* Without major medical problems
* No previous stroke history
* Adequate stability to walk when healthy arm is immobilized
* Active 20 degrees wrist extension and 10 degrees interphalangeal and metacarpophalangeal extension (these movements should be repeated 3 times in 1 minute)

Exclusion Criteria:

* Bilateral stroke or brainstem affected
* Active 20-degree wrist extension and 10-degree interphalangeal and metacarpophalangeal extension
* Global aphasia or cognitive disorders that may affect understanding of test instructions
* Patients with major medical problems that may affect participation
* Existence of neglect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-11-21 (Estimated); Study Completion 2019-11-21 (Estimated)

PRIMARY OUTCOMES:
Motor Activity Log | Patients were examined at baseline
  Motor Activity Log is developed to determine the frequency and quality of use of the affected arm It consists of two scales that question how often the affected side's upper extremity is used for each activity during the 28-day activity (Usage Quantity Scale) and how well it can perform the activity if it uses it. On both scales, the patient scores between 0-5. The score that can be obtained is between 0-5 points and the high score indicates good frequency of use and good quality of movement.
Motor Activity Log | Patients were examined 2 weeks after baseline
  Motor Activity Log is developed to determine the frequency and quality of use of the affected arm It consists of two scales that question how often the affected side's upper extremity is used for each activity during the 28-day activity (Usage Quantity Scale) and how well it can perform the activity if it uses it. On both scales, the patient scores between 0-5. The score that can be obtained is between 0-5 points and the high score indicates good frequency of use and good quality of movement.
Motor Activity Log | Patients were examined 3 months after baseline
  Motor Activity Log is developed to determine the frequency and quality of use of the affected arm It consists of two scales that question how often the affected side's upper extremity is used for each activity during the 28-day activity (Usage Quantity Scale) and how well it can perform the activity if it uses it. On both scales, the patient scores between 0-5. The score that can be obtained is between 0-5 points and the high score indicates good frequency of use and good quality of movement.
Fugl-Meyer Motor Assessment Scale | Patients were examined at baseline
  The Fugl-Meyer Motor Rating Scale, which assesses strength, reflexes and coordination, reflects the stages of motor development. In the evaluation, each item is scored over 2 points. In the upper extremity assessment, 53-66 points are considered as full capacity, 48-52 points are defined as capacity, 32-47 points are considered as limited capacity, and 31 points are considered as under-capacity.
Fugl-Meyer Motor Assessment Scale | Patients were examined 2 weeks after baseline
  The Fugl-Meyer Motor Rating Scale, which assesses strength, reflexes and coordination, reflects the stages of motor development. In the evaluation, each item is scored over 2 points. In the upper extremity assessment, 53-66 points are considered as full capacity, 48-52 points are defined as capacity, 32-47 points are considered as limited capacity, and 31 points are considered as under-capacity.
Fugl-Meyer Motor Assessment Scale | Patients were examined 3 months after baseline
  The Fugl-Meyer Motor Rating Scale, which assesses strength, reflexes and coordination, reflects the stages of motor development. In the evaluation, each item is scored over 2 points. In the upper extremity assessment, 53-66 points are considered as full capacity, 48-52 points are defined as capacity, 32-47 points are considered as limited capacity, and 31 points are considered as under-capacity.
Box-Block Test | Patients were examined at baseline
  Box-Block Test
Box-Block Test | Patients were examined 2 weeks after baseline
  Box-Block Test
Box-Block Test | Patients were examined 3 months after baseline
  Box-Block Test
exercise assessment parameters-cubes lined | Patients were examined at baseline
  cubes lined in 30 seconds
exercise assessment parameters-cubes lined | Patients were examined 2 weeks after baseline
  cubes lined in 30 seconds
exercise assessment parameters-cubes lined | Patients were examined 3 months after baseline
  cubes lined in 30 seconds
exercise assessment parameters-card turned | Patients were examined at baseline
  card turned in 30 seconds
exercise assessment parameters-card turned | Patients were examined 2 weeks after baseline
  card turned in 30 seconds
exercise assessment parameters-card turned | Patients were examined 3 months after baseline
  card turned in 30 seconds
exercise assessment parameters-object gripped | Patients were examined at baseline
  object gripped in 30 seconds
exercise assessment parameters-object gripped | Patients were examined 2 weeks after baseline
  object gripped in 30 seconds
exercise assessment parameters-object gripped | Patients were examined 3 months after baseline
  object gripped in 30 seconds
exercise assessment parameters-water | Patients were examined at baseline
  time it takes to grip and carry a water filled glass to their mouth and putting it back
exercise assessment parameters-water | Patients were examined 2 weeks after baseline
  time it takes to grip and carry a water filled glass to their mouth and putting it back
exercise assessment parameters-water | Patients were examined 3 months after baseline
  time it takes to grip and carry a water filled glass to their mouth and putting it back

SECONDARY OUTCOMES:
Stroke Impact Scale | Patients were examined at baseline
  Stroke Impact Scale 3,0; The aim of the study is to evaluate the perception of the quality of life after stroke by the patients themselves or their caregivers. It is a stroke-specific, patient-centered quality of life measure. It consists of 8 subsections and 59 questions. Each question is scored by evaluating the difficulty experienced in the last week on a 5-point scale. It also includes the assessment of post-stroke recovery perception with a visual analog scale of 0-100 points (0: no improvement, 100: complete recovery)
Stroke Impact Scale | Patients were examined 2 weeks after baseline
  Stroke Impact Scale 3,0; The aim of the study is to evaluate the perception of the quality of life after stroke by the patients themselves or their caregivers. It is a stroke-specific, patient-centered quality of life measure. It consists of 8 subsections and 59 questions. Each question is scored by evaluating the difficulty experienced in the last week on a 5-point scale. It also includes the assessment of post-stroke recovery perception with a visual analog scale of 0-100 points (0: no improvement, 100: complete recovery)
Stroke Impact Scale | Patients were examined 3 months after baseline
  Stroke Impact Scale 3,0; The aim of the study is to evaluate the perception of the quality of life after stroke by the patients themselves or their caregivers. It is a stroke-specific, patient-centered quality of life measure. It consists of 8 subsections and 59 questions. Each question is scored by evaluating the difficulty experienced in the last week on a 5-point scale. It also includes the assessment of post-stroke recovery perception with a visual analog scale of 0-100 points (0: no improvement, 100: complete recovery)

CONTACTS AND LOCATIONS:
Overall Officials: ayşe yalıman, professor, Study Director — istanbul university physical medicine and rehabilitation
Locations (1):
- Istanbul University Istanbul Medicine Faculty, Istanbul, Physical Medicine and Rehabilitation, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yadav RK, Sharma R, Borah D, Kothari SY. Efficacy of Modified Constraint Induced Movement Therapy in the Treatment of Hemiparetic Upper Limb in Stroke Patients: A Randomized Controlled Trial. J Clin Diagn Res. 2016 Nov;10(11):YC01-YC05. doi: 10.7860/JCDR/2016/23468.8899. Epub 2016 Nov 1. PMID 28050492